CLINICAL TRIAL: NCT01766830
Title: Evaluation of Rapid Diagnostic Tests (RDT) in Association With Clinical and Laboratory Predictors for the Diagnosis of Neglected Tropical Diseases (NTD) in Patients Presenting With Persistent Fever (≥1 Week) in Cambodia, Nepal, Democratic Republic of the Congo and Sudan
Brief Title: Rapid Diagnostic Tests and Clinical/Laboratory Predictors of Tropical Diseases In Patients With Persistent Fever in Cambodia, Nepal, Democratic Republic of the Congo and Sudan (NIDIAG-Fever)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); B.P. Koirala Institute of Health Sciences (Other); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); University of Khartoum (Other); Sihanouk Hospital Center of HOPE (Other)
Responsible Party: Principal Investigator, Francois CHAPPUIS, Professor, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WP2-01-FEV; 260260 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Visceral Leishmaniasis; Human African Trypanosomiasis; Enteric Fever; Melioidosis; Brucellosis; Leptospirosis; Relapsing Fever; Rickettsial Diseases; HIV; Tuberculosis; Malaria; Amoebic Liver Abscess
MeSH Terms: conditions — Leishmaniasis, Visceral; Typhoid Fever; Melioidosis; Brucellosis; Leptospirosis; Relapsing Fever; Rickettsia Infections; Tuberculosis; Malaria; Liver Abscess, Amebic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 3 Diagnostic (Experimental): A total of 10 RDTs will be assessed in the patients cohort for the respective target condition
  Interventions: Device: rk28 ICT; Device: IT LEISH (rK39); Device: Immunochromatographic HAT test; Device: HAT Serostrip; Device: Card Agglutination Trypanosoma Test (CATT)-10; Device: Typhidot M; Device: S. typhi IgM/IgG; Device: Test-it Typhoid IgM; Device: Test-it Leptospirosis IgM; Device: Leptospira IgG/IgM

INTERVENTIONS:
Device: rk28 ICT — rk28 ICT is an immunochromatographic assay intended for qualitative detection of IgG antibodies directed towards VL in human serum, plasma or whole blood. It is manufactured by EASE-Medtrend (Shanghai, China)
Device: IT LEISH (rK39) — IT LEISH is an immuno-chromatographic test, using the recombinant antigen K39, to detect the presence of antibodies against Leishmania spp. It is manufactured by BioRad laboratories, USA.
Device: Immunochromatographic HAT test — This is a lateral flow immunochromatographic test manufactured by Standard Diagnostics (Korea) in collaboration with FIND.
Device: HAT Serostrip — The HAT Serostrip is an immunochromatographic assay developed by Coris BioConcept, France, which is designed for remote field use in individual HAT suspects.
Device: Card Agglutination Trypanosoma Test (CATT)-10 — The Card Agglutination Trypanosoma test (CATT) has been used for many years at large scale for mass screening of mostly asymptomatic individuals (CATT-R250). Unfortunately, its operating characteristics have only been evaluated in the context of patients with persistent fever. Although it is not strictly an RDT, the CATT is rather easily performed in remote settings, in particular since a new and more robust format (CATT-D10) allows to test a lower number of patients in peripheral health facilities. It is manufactured by the Institute of Tropical Medicine of Antwerp, Belgium.
Device: Typhidot M — The Typhidot M test is a dot enzyme immunoassay that detects IgM and IgG directed against Salmonella typhi. It is manufactured by Reszon Diagnostics International, Malaysia
Device: S. typhi IgM/IgG — The Salmonella typhi IgG/IgM Rapid Test is an immunochromatographic assay for the qualitative differential detection of IgG and IgM antibodies to Salmonella typhi in human serum, plasma or whole blood. It is manufactured by Standard Diagnostics (Korea)
Device: Test-it Typhoid IgM — Test-it Typhoid IgM lateral flow assay is a one-step immunochromatographic assay which uses a lipopolysaccharide (LPS) antigen derived from salmonella typhi for the detection of specific IgM antibodies. It is manufactured by Life Assay, South Africa.
Device: Test-it Leptospirosis IgM — The Test-it™ Leptospira lateral flow device detects IgM antibodies in humans against Leptospira in whole blood or serum. It is manufactured by Life Assay, South Africa
Device: Leptospira IgG/IgM — This test enables the differential detection of IgG and IgM antibodies to Leptospira interrogans. It is manufactured by Standard Diagnostics, Korea

SUMMARY:
Tropical fevers have been a diagnostic challenge from the antiquity. Nowadays, despite the availability of good diagnostic capacities, undifferentiated febrile illnesses continue to be a thorny problem for travel physicians. In developing countries, the scarcity of skilled personnel and adequate laboratory facilities makes the differential diagnosis of fevers even more complex. Health care workers must often rely on syndrome-oriented empirical approaches to treatment and might overestimate or underestimate the likelihood of certain diseases. For instance Neglected Tropical Diseases (NTD) contribute substantially to the burden of persistent (more than 1 week) fevers in the Tropics, causing considerable mortality and major disability. These diseases are however rarely diagnosed at primary health care (PHC) level. The difficulty in establishing the cause of febrile illnesses has resulted in omission or delays in treatment, irrational prescriptions with polytherapy, increasing cost and development of drug resistance.

In resource-limited settings, clinical algorithms constitute a valuable aid to health workers, as they facilitate the therapeutic decision in the absence of good laboratory capacities. There is a critical lack of appropriate diagnostic tools to guide treatment of NTDs. While clinical algorithms have been developed for some NTDs, in most cases they remain empirical. Besides, they rarely take into account local prevalence data, do not adequately represent the spectrum of patients and differential diagnosis at the primary care level and often have not been properly validated. The purpose of the study is to develop evidence-based Rapid Diagnostic Test (RDT)-supported diagnostic guidelines for patients with persistent fever (≥ 1 week) in the Democratic Republic of the Congo (DRC), Sudan, Cambodia and Nepal.

DETAILED DESCRIPTION:
This study is part of a large European Union (EU)-funded research project called NIDIAG that aims at developing integrated, evidence-based syndromic approach to improve management of NTD-related clinical syndromes. NIDIAG targets three non-specific clinical syndromes: the persistent fever, neurological, and intestinal syndrome. The objective of the project is to establish diagnostic guidelines for each of this syndrome, with a particular focus on severe and treatable neglected infectious diseases. The developed guidelines should integrate relevant Point-of-Care (POC)tests.

The persistent fever syndrome targeted by NIDIAG is defined as presence of fever for at least one week. The list of diseases - both NTD and other Infectious Diseases (ID) - that frequently cause persistent (≥1 week) fever in the study countries includes: Visceral Leishmaniasis (VL), Human Africa Trypanosomiasis (HAT), Enteric (typhoid, paratyphoid) fever, Malaria, Brucellosis, Melioidosis, Tuberculosis, Amoebic liver abscess, Relapsing fever, HIV, Rickettsial diseases, and Leptospirosis. The study will try to identify clinical and laboratory predictors of these diseases as well as validate existing RDTs.

ELIGIBILITY:
Inclusion Criteria:

* fever for ≥ 1 week
* ≥ 5 years old (18 years onward in Cambodia)

Exclusion Criteria:

* unwilling or unable to give written informed consent
* unable in the study physician's opinion to comply with the study requirements
* existing laboratory confirmed diagnosis
* need of immediate intensive care due to shock or respiratory distress

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1927 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of Visceral Leishmaniasis (VL), Human African Trypanosomiasis (HAT) and other Neglected Tropical Diseases (NTDs) | 18 months
  Number of patients diagnosed with VL, HAT and other NTDs among those presenting with persistent(≥ 1 week) fever in one of the study sites
Identification of clinical and laboratory diagnostic indicators | 18 months
  Sensitivity, specificity, crude and adjusted likelihoods ratios (LR), and predictive values (post-test probabilities) of clinical and first-line laboratory predictors for the diagnosis of VL, HAT and other NTDs
Identification of reliable Rapid Diagnostic Tests (RDTs) | 18 months
  Assessment of sensitivity, likelihood ratios and performances (diagnostic accuracy) of the novel study RDTs for VL, HAT, enteric fever and
Predictive values of RDTs | 18 months
  Predictive values (post-test probabilities) of RDTs, alone and in combination, for the respective target conditions within the multi-disease approach

SECONDARY OUTCOMES:
Cost-effectiveness of the diagnostic tests | 18 months
  Unit costs of diagnostic tests for the diagnosis of HAT and other priority NTDs/IDs in the setting

CONTACTS AND LOCATIONS:
Overall Officials: François Chappuis, MD, PhD, Study Director — University Hospital, Geneva
Locations (7):
- Sihanouk Hospital Center of HOPE, Phnom Penh, Cambodia
- Democratic Republic of the Congo (2):
  - Reference Hospital Mosango and Kasay Health Centre, Mosango, Bandundu
  - Institut National de Recherche Biomédicale, Kinshasa
- Nepal (2):
  - Dhankuta District hospital, Dhankutā, Koshi Zone
  - BP Koirala Institute of Health Sciences, Dharān
- Sudan (2):
  - Tabarak Allah Hospital, Tabarak Allah, Al Qaḑārif
  - University of Khartoum, Khartoum

REFERENCES:
- [Derived] Bottieau E, Van Duffel L, El Safi S, Koirala KD, Khanal B, Rijal S, Bhattarai NR, Phe T, Lim K, Mukendi D, Kalo JL, Lutumba P, Barbe B, Jacobs J, Van Esbroeck M, Foque N, Tsoumanis A, Parola P, Yansouni CP, Boelaert M, Verdonck K, Chappuis F. Etiological spectrum of persistent fever in the tropics and predictors of ubiquitous infections: a prospective four-country study with pooled analysis. BMC Med. 2022 May 2;20(1):144. doi: 10.1186/s12916-022-02347-8. PMID 35491421
- [Derived] Alirol E, Horie NS, Barbe B, Lejon V, Verdonck K, Gillet P, Jacobs J, Buscher P, Kanal B, Bhattarai NR, El Safi S, Phe T, Lim K, Leng L, Lutumba P, Mukendi D, Bottieau E, Boelaert M, Rijal S, Chappuis F. Diagnosis of Persistent Fever in the Tropics: Set of Standard Operating Procedures Used in the NIDIAG Febrile Syndrome Study. PLoS Negl Trop Dis. 2016 Nov 3;10(11):e0004749. doi: 10.1371/journal.pntd.0004749. eCollection 2016 Nov. PMID 27812090
- See also: NIDIAG Consortium website — http://www.nidiag.org/